CLINICAL TRIAL: NCT05247515
Title: Evaluation of Nexpowder Application to Prevent Delayed Bleeding After Large Colorectal Endoscopic Mucosal Resection
Brief Title: Evaluation of Nexpowder Application to Prevent Delayed Bleeding After Colorectal Endoscopic Mucosal Resection
Acronym: NEXBLEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gabriel RAHMI (Other)
Responsible Party: Sponsor-Investigator, Gabriel RAHMI, Principal Investagator, Medical Doctor, French Society of Digestive Endoscopy
Organization: French Society of Digestive Endoscopy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFED 154
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal polypectomy; endoscopic mucosal resection; hemostatic powder
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group: Nexpowder application on the scar after EMR with coagulation of visible vessels (Experimental): To compare of the risk of bleeding after EMR application of nexpower (not a drug but a device with CE mark) on the resect area (scar) to cover the whole surface of mucosal resection.
  Interventions: Device: Endoscopic mucosal resection with nexpowder
- standard procedure : EMR with coagulation of visible vessels (No Intervention): After EMR with coagulation of visible vessels, if the patient is randomized in the comparative group, not nexpowder will be applied on the scar (common practice)

INTERVENTIONS:
Device: Endoscopic mucosal resection with nexpowder — At the end of the EMR procedure, the patient will be randomized. In the treated group, Nexpowder will be sprayed thanks to a catheter inserted through the operating channel of the endoscope.
  Arms: Treated group: Nexpowder application on the scar after EMR with coagulation of visible vessels

SUMMARY:
Delayed bleeding is the most frequent (5 to 15%) and challenging complication after large colorectal polypectomy. Different preventive treatments, such as the prophylactic use of clips, have been tried to prevent the occurrence of delayed bleeding, but to date, no treatment has clearly shown its effectiveness. In addition, preventive hemostasis with clips is difficult and costly. A newly developed endoscopic hemostatic powder generating gelation effect (Nexpowder) may be an effective alternative to prevent post polypectomy bleeding in patients treated by endoscopic mucosal resection (EMR) for large superficial colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Indication of EMR for a superficial nonpedunculated colorectal lesion
* Higher risk of bleeding (score GSEED RE2 ≥ 7*)

  *Score GSEED RE2 (Albeniz et al GIE 2020):
* Proximal location (cecum to transverse included) : 3 points
* Antiplatelets or anticoagulation use: 3 points
* Lesion size ≥ 40 mm: 1 point
* ASA III-IV or major comorbidity: 1 point

Exclusion Criteria:

* Patients susceptible to allergic reactions to certain substances in Nexpowder
* More than one colorectal lesion
* Suspicion of invasive cancer (Kudo V, Sano IIIb, Connect III), macronodular more than 1 cm, depressed area (Paris IIc)
* Pedunculated polyps (Ip from Paris classification) or ulcerated polyps (III)
* Recurrent or residual lesion after endoscopic or surgical resection
* Poor bowel preparation quality (Boston score < 6)
* Inflammatory bowel disease (IBD)
* Patients with a platelet count of 50,000/mm3 or less
* Patients with acquired (non-medicated) or inherited bleeding disorders
* Patients with advanced cancer or inflammatory bowel disease, including ulcerative colitis (with colonic involvement)
* Contraindication to general anesthesia
* Women who are pregnant or who wish to become pregnant during the study or women who are breastfeeding.
* Children, immunocompromised persons and persons over 90 years of age
* Patients already participating or scheduled to participate in other clinical trials
* Lesion previously resected by endoscopy
* Patient with an initial metastatic lesion before colonoscopy
* Patient unable to give personal consent
* Lack of signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Severe post-resection bleeding rate up to Day 30 | 30 days
  Number of patients with a severe post-resection bleeding. It is defined as bleeding requiring a new endoscopy or surgery, OR a radiological embolization, OR blood transfusion, OR a re-hospitalization OR haematochezia with hemoglobin loss > 2 g/dl

SECONDARY OUTCOMES:
The success rate of Nexpowder application | Day of resection
  Number of patients with a satisfactory covering of the scar by the powder
Delayed perforation rate | 30 days
  Number of patients with a presence of air and fluid into the peritoneal cavity on the CT scanner
Stenosis rate | 30 days
  Number of patients with the impossibility to pass through the lumen with a standard colonoscope
Post coagulation syndrome | 30 days
  Number of patients with a fever and abdominal pain without air or fluid into the peritoneal cavity on the CT scanner.
Bowel obstruction rate | 30 days
  Number of patients with at least one symptomatic bowel obstruction.
Rate of cases requiring transfusion related to post-EMR bleeding | 30 days
  Number of patients for whom at least one transfusion was ordered after the EMR
Rate and duration of hospitalizations | 30 days
  Number of hospitalizations and number of days of hospitalization per stay within 30 days after EMR

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Européen Georges Pompidou, 20 Rue Leblanc, Paris, France